CLINICAL TRIAL: NCT03841279
Title: Utilizing MRI for Earlier Diagnosis of Rheumatoid Arthritis
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kerry Wright, Principal Investigator, Mayo Clinic
Other Study IDs: 18-005455
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: MRI — Magnetic resonance imaging (MRI) produces detailed images of the body's internal structures without relying on radiation. It is used to diagnose and also gauge efficacy of treatment.

SUMMARY:
MRI has been shown to be helpful in identifying patients who present with undifferentiated inflammatory arthritis who will develop RA within a one year follow up period. The absence of other clinically apparent symptoms often causes delays in diagnosis of RA. The use of the MRI in conjunction with the physical examination has the potential to reduce diagnostic delay. Earlier diagnosis would allow for earlier treatment implementation for better patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

≥ 18 years old

Undifferentiated inflammatory arthritis suspected to be early RA (≥1 joint with synovitis and ≥1 other tender joint)

Symptom duration ≤1 year

Exclusion Criteria:

Unwillingness or inability to return to Mayo Clinic Rochester for research follow-up visits

Current or previous use of DMARDS

Taking ≥10 mg of prednisone a day

Contraindications to contract enhanced MRI

History of another definite autoimmune or inflammatory rheumatic disease

History of psoriasis

History of inflammatory bowel disease

Unsuitably as deemed by the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study will be patients with undifferentiated inflammatory arthritis or seronegative rheumatoid arthritis from the outpatient practice of the Division of Rheumatology in Rochester, MN.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Earlier Diagnosis of RA if MRI is utilized | 1 year
  To determine if MRI is predictive of later development of RA in patients with undifferentiated inflammatory arthritis; patients with inflammatory arthritis who receive an MRI will have earlier initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Wright, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No